CLINICAL TRIAL: NCT03509519
Title: Impact of Neuromuscular Electrical Stimulation on Physical Function in Older Adults
Brief Title: Neuromuscular Electrical Stimulation and Physical Function in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas State University (Other)
Responsible Party: Principal Investigator, Joni Mettler, Assistant Professor, Texas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REPFY18
Record Dates: First submitted 2018-03-07; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Sarcopenia
Keywords: neuromuscular electrical stimulation; physical activity; muscular strength
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This clinical trial will use a pre-test - post-test randomized experimental design. Subject will be randomly assigned to the treatment group or the sham group. Study outcomes will be measured pre- and post-intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES-Millicurrent Group (Experimental): NMES-millicurrent group will receive the NMES experimental treatment. Stimulating electrodes will be applied to the quadriceps muscle of each leg 3 times a week for 4 weeks (12 sessions) for 40min on each leg.
  Interventions: Other: NMES-Millicurrent
- NMES-Microcurrent Group (Sham Comparator): The NMES-microcurrent group will receive the Sham Treatment. The Sham Treatment will consist of electrode pad application for 40 mins on each leg, but electrical current will not be delivered. Otherwise all procedures will be the same as the NMES-millicurrent experimental group. Participants will be informed they are receiving microcurrent stimulation which is typically not felt by patients. Microcurrent stimulation is an actual type of electrical stimulation that is used therapeutically and is typically not felt by patients, however, participants will not receive this treatment. Participants will be informed of the actual treatment received at the study conclusion. Those in the Sham Group will be given the opportunity to receive the treatment at the conclusion of the study.
  Interventions: Other: NMES-Millicurrent

INTERVENTIONS:
Other: NMES-Millicurrent — Stimulating electrodes will be applied to the quadriceps muscle of each leg 3 times a week for 4 weeks (12 sessions) for 40min per leg.

SUMMARY:
The purpose of this placebo controlled clinical trial is to examine the effects of of neuromuscular electrical stimulation (NMES) training on physical activity, muscle function, self-efficacy, and blood markers [e.g., brain-derived neurotrophic factor (BDNF)] in older adults.

It is hypothesized that 4-weeks of NMES will increase 1) physical activity, 2) muscle function, 3) self-efficacy, and 4) BDNF in older adults.

Sarcopenia is a destructive progressive cycle of impaired physical function resulting in loss of muscle mass, strength, and self-confidence in ability to perform physical activities, compounded by difficulty walking and ultimately reduced physical activity levels for many older adults. Neuromuscular electrical stimulation (NMES) is a common therapeutic modality used to create involuntary muscle contractions as a means to increase muscle strength, and may be an effective treatment for improving muscle function and physical activity levels in older adults with sarcopenia. Thus, it is critical to explore viable and effective alternative therapies to increase physical activity. The goal of the investigators' is to determine the effectiveness of neuromuscular electrical stimulation (NMES) at increasing physical activity and related biological, psychological, and muscle function factors. This placebo controlled clinical trial will use a pre-test - post-test randomized experimental design.

DETAILED DESCRIPTION:
Older healthy adults (60 and older) will participate in this study. Participants will undergo 4 weeks of neuromuscular electrical stimulation (NMES) training. Participants will be randomized into the one of two groups 1) NMES-millicurrent or 2) NMES microcurrent. Participants will undergo pre- and post-training testing for muscle function, physical function, and psychological variables related to physical activity. Blood samples will also be obtained pre- and post-training.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy men and women
* ages 60 and older

Exclusion Criteria:

* 1) they have participated in regular resistance training exercise or physical rehabilitation of the lower extremity within 2 months of the study
* 2) contraindicating conditions for electrical stimulation are present (i.e., swollen, infected or inflamed areas including open wounds, or painful areas on the lower limbs, implanted electronics including cardiac pacemakers, electronic infusion pumps, implanted stimulators, or surgical hardware in the lower limbs)
* 3) they have current knee injury or knee pain
* 4) have a neuromuscular disease
* 5) currently taking insulin for diabetes regulation
* 6) they have a history of seizures

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity | Physical activity levels will be assessed for 1 week before the intervention and for 1 week after the intervention period. The change in physical activity will be compared between these two time-periods.
  Physical activity will be measured from accelerometer data.

SECONDARY OUTCOMES:
Change in Muscle Strength | Muscle strength will be assessed prior to the first day of the intervention, after 2-weeks of the intervention, and two days after the completion of the 4-week intervention.
  Muscle strength will be measured by maximal voluntary contraction on a dynamometer.
Change in Muscle Endurance | Muscle endurance will be assessed prior to the first day of the intervention and 2 days after the completion of the 4-week intervention.
  Muscle endurance time will be measured on a dynamometer.
Pre-training NMES-related change in glucose | Blood glucose will be measured immediately before and immediately after the application of the intervention on the first (training Day 1) NMES intervention day.
  Fasting blood glucose levels will be measured.
Post-training NMES-related change in glucose | Blood glucose will be measured immediately before and immediately after the application of the intervention on the last day (training day 12) of the NMES intervention.
  Fasting blood glucose levels will be measured.
Pre-training NMES-related change in Brain-derived Neurotrophic Factor (BDNF) levels | BDNF levels will be measured immediately before and immediately after the application of the intervention on the first (training Day 1) NMES intervention day.
  Brain-derived neurotrophic factor, a marker of neuronal growth, will be obtained from a blood sample.
Post-intervention change in Brain-derived Neurotrophic Factor (BDNF) levels | BDNF levels will be measured immediately before and immediately after the application of the intervention on the last day (training day 12) of the NMES intervention.
  Brain-derived neurotrophic factor, a marker of neuronal growth, will be obtained from a blood sample.
Change in self-efficacy of activities of daily living | Self-efficacy will be measured prior to the first day of the intervention and 4 days after the last day of the 4-week intervention.
  Self-efficacy will be measured by survey.
Change in motor activation | Motor activation will be measured prior to the first day of the intervention and two days after the completion of the 4-week intervention.
  Motor activation will be measured by surface electromyography measures.
Change in perception of pain | Perceptions of pain will be measured immediately after the NMES treatment on the first (training day 1) and last day (training day 12) of the 4-week intervention.
  Perceived pain experienced during the NMES treatment will be measured by survey.
Physical activity during the 4-week intervention | Physical activity levels will be measured during the 4 weeks of the intervention (from the first day of the intervention through the last day of the intervention).
  Physical activity will be measured from accelerometer data.
Change in timed up and go test | Timed up and go test will be assessed prior to the first day of the intervention and 4 days after the last day of the 4-week intervention.
  The timed up and go test will measure the time it takes to stand up from a chair, walk a few meters, turn around and sit back down.
Change in stair climb test | The stair cimb test test will be assessed prior to the first day of the intervention and 4 days after the last day of the 4-week intervention.
  The stair climb test will assess the time it takes to safely ascend 10 stairs.
Change in five repetition sit-to-stand test | The five repetition sit-to-stand test will be assessed prior to the first day of the intervention and 4 days after the last day of the 4-week intervention.
  The five repetition sit-to-stand test will assess the time it take to stand up and sit down on a chair 5 times.
Change in 6-min walk test | The 6-min walk test will be assessed prior to the first day of the intervention and 4 days after the last day of the 4-week intervention.
  The 6-min walk test will assess the distance an individual can walk in 6 minutes.
Change in grip strength | The grip strength test will be assessed prior to the first day of the intervention and 4 days after the last day of the 4-week intervention.
  The grip strength test will measure the maximal hand grip strength of both hand using a grip strength dynamometer.
Change in arm curl test | The arm curl test will be assessed prior to the first day of the intervention and 4 days after the last day of the 4-week intervention.
  The arm curl test will measure the number of repetitions completed with a dumbbell.

CONTACTS AND LOCATIONS:
Overall Officials: Joni A Mettler, PhD, Principal Investigator — Texas State University

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data with other researches until the data are published in journals and presented at conferences.

REFERENCES:
- [Background] Kemmler W, von Stengel S, Engelke K, Haberle L, Kalender WA. Exercise effects on bone mineral density, falls, coronary risk factors, and health care costs in older women: the randomized controlled senior fitness and prevention (SEFIP) study. Arch Intern Med. 2010 Jan 25;170(2):179-85. doi: 10.1001/archinternmed.2009.499. PMID 20101013
- [Background] Kern H, Barberi L, Lofler S, Sbardella S, Burggraf S, Fruhmann H, Carraro U, Mosole S, Sarabon N, Vogelauer M, Mayr W, Krenn M, Cvecka J, Romanello V, Pietrangelo L, Protasi F, Sandri M, Zampieri S, Musaro A. Electrical stimulation counteracts muscle decline in seniors. Front Aging Neurosci. 2014 Jul 24;6:189. doi: 10.3389/fnagi.2014.00189. eCollection 2014. PMID 25104935
- [Background] Janssen I, Shepard DS, Katzmarzyk PT, Roubenoff R. The healthcare costs of sarcopenia in the United States. J Am Geriatr Soc. 2004 Jan;52(1):80-5. doi: 10.1111/j.1532-5415.2004.52014.x. PMID 14687319